CLINICAL TRIAL: NCT01161797
Title: Correlation Between 1,5-anhydroglucitol and Postprandial Hyperglycemia by Continuous Glucose Monitoring System and Clinical Usefulness of 1,5-anhydroglucitol in Well-controlled Diabetic Patients
Brief Title: 1,5-AG as a Marker of Postprandial Hyperglycemia and Glucose Variability in Well-controlled Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Jeong-taek Woo, MD, PhD, Kyunghee University Medical Center
Other Study IDs: KMC-ENDO-0801
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: 1,5-Anhydroglucitol
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum (HbA1c, fructosamine, 1,5-anhydroglucitol)
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study was to evaluate the correlation between 1,5-Anhydroglucitol in patients with HbA1C <7%, and glycemic excursions as assessed by the continuous glucose monitoring system compared to fructosamine.

DETAILED DESCRIPTION:
1,5-Anhydroglucitol (AG) is a glucose analogue present in the plasma of healthy subjects. Physiologically, the plasma levels of 1,5-AG are very stable and only a small quantity is excreted in the urine. It is competitively reabsorbed with glucose in the renal tubules. Therefore, in the hyperglycemic state where glycosuria is present, glucose competitively inhibits renal tubular reabsorption of 1,5-AG and consequently the plasma 1,5-AG levels decrease. When glycemia is normalized and glycosuria is resolved, 1,5-AG levels increase.

The usefulness of 1, 5-AG in reflecting glycemic excursions have been demonstrated in moderately controlled patients to some extent, although some studies reveal controversial results.

Therefore, the aim of this study was to evaluate the association of 1,5-AG and postprandial hyperglycemia determined using the Continuous Glucose Monitoring System (CGMS) in DM patients with HbA1C<7% and evaluate the usefulness of 1,5-AG as a marker of glycemic control compared to HbA1C and fructosamine.

ELIGIBILITY:
Inclusion Criteria:

* HbA1C < 7%
* HbA1c modification <0.5% in the previous 3 months
* no recent addition of oral hypoglycemic medications or change in insulin dose >10% previous 3 months

Exclusion Criteria:

* pregnancy
* anemia (Hb <10.0 g/dL)
* liver disease (ALT >2 UNL)
* hypoalbuminemia (albumin <3.5 g/dL)
* serum creatinine >2 mg/dL
* acute or chronic renal tubulointerstitial disease
* severe medical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Well-controlled patients with type 2 diabetes with HbA1c<7%
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2008-02; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
postprandial hyperglycemia | 3days
glucose variability | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-taek Woo, MD, PhD, Study Director — Department of Endocrinology and Metabolism, Kyung Hee University School of Medicine, Seoul, Korea
Locations (1):
- Kyunghee University Medical Center, Seoul, South Korea